CLINICAL TRIAL: NCT06678035
Title: Use of Simplified Lung Ultrasound Score for Predicting ICU Outcomes in Patients with Acute Respiratory Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Zakaria Hassab Elnabi Shahin, Resident doctor Principal investigator, Assiut University
Other Study IDs: Chest US in ICU
Record Dates: First submitted 2024-10-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Pneumnia; Chest Infection; Critically-ill Patients Admitted to the ICU for Acute Respitatory Failure, Regardless the Aetilogy
Keywords: LUS; Acute respiratory failure; Critically-ill patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to

Primary Aims:

Verify the predictability of the PLIS at admission in predicting major clinical outcomes including:

* ICU mortality (or discharge) and time to death (or discharge)
* Escalation of ventilatory support antibiotic therapy or supportive medications (inotropes, steroids, sedation, neuromuscular blockers).

Secondary Aims:

* Determine the correlation between initial PLIS and the degree of disease severity (as evaluated per SOFA and APACHE II scores)
* Determine the correlation between initial PLIS and partial pressure of oxygen in arterial blood (PaO2) to Fraction of inspired oxygen (FiO2): PaO2/FiO2
* Explore the potential association between the type of ventilatory support, ventilatory settings and PLIS at different time points.
* Verify whether the site of consolidation (anterior vs. posterior lung zones) can reliably predict mortality in in ALI patients.
* Determine the correlation between the PLIS score and the degree of ALI as quantified by CT of the chest (whenever a CT study is available) at the time of admission.

DETAILED DESCRIPTION:
Respiratory failure and acute lung injury (ALI) in patients admitted to ICU are major causes of morbidity And mortality As high as 60 % of ICU population dii during their ICU admission due to ALI Accurate assessment of the severity of ALI is Crucial for guiding treatment decisions and predicting patient outcome Reliance on chest X-ray and Computed tomography has its limitations including subjectivity and potential delays in obtaining and interpreting results high cost radiation exposure and lack of continuous monitoring particularly for critically ill patients Ultrasound -being non-invasive low cost radiation free- has been increasingly used as a bedside tool for evaluation and monitoring of ALI However most lung ultrasound protocols published to date are cumbersome and time consuming They typically involve screening at least 12 different lung areas each graded from 0 to 3 point thus generating scores ranging from 0 to 36 .While these scores are informative for research purposes they are less practical in a busy or ICU environment Also disregarding the site of B-lines or consolidation and the size of consolidation potentially under-estimates the severity of ALI Recently a novel -yet comprehensive- point of care ultrasound lung injury score has been developed to aid informative and quick assessment of ALI in ICU PLIS involves screening of only 3 areas but it uniquely considers the level of ventilatory support and gives credit to the number of B lines size of consolidation location of consultation The score reliably predicted to the need of ICU admission in a group off of COVID 19 patients directly correlation with their SOFA scores also predicted ICU mortality in this patient However Wider adoption of PLIS by intensivists dictates evaluation of its performance in a wider ICU population with a variety of underlying diagnoses This study is to verify whether PLIS remains valid for predicting ICU outcomes in patients with acute respiratory failure regardless the etiology type of respiratory failure oxygen requirement level of ventilatory support

ELIGIBILITY:
Inclusion Criteria:

* Age is or more than 18 years old.
* Admission to ICU in the first24 hours at time of recruitment to the study.
* Patients in respiratory failure [PaO2 is less then 60 % mmHg]

Exclusion Criteria:

* Co- existing chronic lung disease, pathology of which is known display abnormalities on US examination (interstitial lung diseases, bronchiectasis).
* Large pneumothorax or massive pleural effusion causing significant collapse and precluding proper visualization of underlying lung.
* Conditions that may interfere with lung ultrasound quality or probe contact such as marked obesity, severe chest wall deformities, burns or wounds.

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are more than 18 years in repiratory failure in ICU and use of chest us in supine or semisupine position
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
ICU Mortality | 60 days
  Percentage of patients who will die during their ICU admission
Time to death/discharge | 60 days
  Number of days until the patient dies inside the ICU or becomes discharged from ICU

SECONDARY OUTCOMES:
Need for Therapy escalation: Ventilatory Support | 60 days
  Binary response (yes or no), to whether the type of ventilatory support (COT-HVNI-NIV-IMV) was escalated or not
Need for Therapy Escalation: Ventilatory seetings | 60 days
  Binary response (yes or no) to whether change in ventilatory settings (FiO2, IPAP, EPAP, Ti,TVe) was needed
Need for Therapy Escalation: Medications | 60 days
  Binary response (yes/no) to whether medications like antibiotics, inotropes, sedation, or NMBs, which were not initiated needed to be added or not

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marchioni A, Castaniere I, Tonelli R, Fantini R, Fontana M, Tabbi L, Viani A, Giaroni F, Ruggieri V, Cerri S, Clini E. Ultrasound-assessed diaphragmatic impairment is a predictor of outcomes in patients with acute exacerbation of chronic obstructive pulmonary disease undergoing noninvasive ventilation. Crit Care. 2018 Apr 27;22(1):109. doi: 10.1186/s13054-018-2033-x. PMID 29703214
- [Background] Biasucci DG, Buonsenso D, Piano A, Bonadia N, Vargas J, Settanni D, Bocci MG, Grieco DL, Carnicelli A, Scoppettuolo G, Eleuteri D, DE Pascale G, Pennisi MA, Franceschi F, Antonelli M; Gemelli Against COVID-19 Group. Lung ultrasound predicts non-invasive ventilation outcome in COVID-19 acute respiratory failure: a pilot study. Minerva Anestesiol. 2021 Sep;87(9):1006-1016. doi: 10.23736/S0375-9393.21.15188-0. Epub 2021 Jul 14. PMID 34263580
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29703214/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34263580/